CLINICAL TRIAL: NCT06078488
Title: Individualized Nutritional Care Bundle for Home Nursing Patients With Pressure Injuries - A Cluster-Randomized, Pragmatic Clinical Trial and Economic Evaluation.
Brief Title: Individualized Nutritional Care Bundle for Home Nursing Patients With Pressure Injuries.
Acronym: INCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: Home Nursing Foundation (HNF) (Unknown); Duke-NUS Graduate Medical School (Other); Temasek Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCA
Record Dates: First submitted 2023-07-31; First posted 2023-10-11 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-10

CONDITIONS: Wounds and Injuries; Malnutrition; Nutritional Deficiency; Wound Healing Delayed; Nurse's Role
Keywords: Pressure Injury; Nutritional Support; Community Nursing; Clinical Nutrition; Malnutrition
MeSH Terms: conditions — Wounds and Injuries; Malnutrition; Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Subjects will not be blinded to group allocations due to the nature of the study, which is not a placebo-controlled trial, but rather, a real-world pragmatic study. Subjects, research dietitian and nursing staff will be aware that they are in a study to examine the effects of nutritional intervention on pressure injury healing rates. The nursing personnel responsible for measuring wounds and gathering data will not be blinded, given their role in conducting follow-up with the participants as a component of clinical care. However, they will be randomized to ensure that they do not attend to both the intervention and control groups. The research dietitian will be blinded to the measurement and health outcomes. The trial statistician will be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Individualized and Protocolized Nutrition Care Bundle with Nutritional Supplementation, Education and Support by Nurses trained in Nutritional Management and Dietitians.
  Interventions: Other: Individualized and Protocolized Nutritional Care Bundle
- Control (Experimental): Nursing Care by Nurses trained in Nutritional Management, with or without Supplements.
  Interventions: Other: Optimized Standard Care

INTERVENTIONS:
Other: Individualized and Protocolized Nutritional Care Bundle — Education on nutritional and wound care for patient/family based on the latest guidelines based on the "The European Pressure Ulcer Advisory Panel, the National Pressure Injury Advisory Panel, and the Pan Pacific Pressure Injury Alliance Prevention and Treatment of Pressure Ulcers/Injuries: 2019 Clinical Practice Guideline". A dietetic consultation at baseline, week 4 and week 8 on optimizing nutritional intake to meet caloric/protein requirements, along with additional high protein high energy (HPHE) supplementation prescribed for those participants who do not meet nutritional requirements (25-35kcal/kg/d and 1.2-2.0g protein/kg/d). The dietetic consultation will be done via face-to-face home visits and/or telehealth. A specialised nutritional supplement containing 4.5 g Arginine, 156 mg Vitamin C, 40.9 mg alpha-tocopherol equivalents (Vitamin E), 30 kcal will be administered twice a day via oral ingestion or tube feeding (mixed in 100ml water) for 12 weeks.
  Arms: Intervention
Other: Optimized Standard Care — Only receiving education and management from specialized nurses trained in nutritional management , with or without supplementation
  Arms: Control

SUMMARY:
Objective:

To evaluate the impact of an individualized nutrition intervention package on pressure injury healing rates, prevention of new pressure injuries, complications, quality of life, and cost-effectiveness in adult on home nursing care with pressure injuries staged II and above in Singapore.

Study Design:

A two-group, non-blinded, randomized, pragmatic clinical trial with a cost-effectiveness analysis.

Location/ Setting:

Community

Participants:

Adults (aged 21 years and above) receiving home nursing care with at least one pressure injury (Stage II, III, IV, or Unstageable).

190 subjects per arm

Intervention:

The intervention group will receive an individualized nutrition intervention package consisting of individualized nutritional supplementation, specialized nutritional education pamphlets, regular dietetic support via home visits or telehealth, and home nursing care by nurses trained in nutrition care.

The control group will receive specialized nutritional educational pamphlets, and home nursing care by nurses trained in nutrition care, with or without nutritional supplementation.

Outcome Measures:

Main outcomes of wound area reduction, and proportion of participants with >40% area reduction at 30 days, 60 days and 90 days. Secondary outcomes include proportion of participants and wounds with increasing severity of PI stages (e.g., stage II to stage III), improvement in Health-Related Quality of Life (HRQOL) and nutritional status, and incidence of wound infections at 30 days, 60 days and 90 days, proportion of participants with complete healing, mortality and unplanned hospital admissions.

Economic Evaluation:

The primary economic outcome will be the incremental cost-effectiveness ratio (ICER) per pressure injury prevented, with a time horizon of 1 year for intervention versus control during the period of intervention (3-months) and up to a year.

Statistical Analyses:

Individual patient level analysis will be performed as per our primary analysis, and we will also perform cluster level analysis. Hazard ratios (HR) will be determined using Cox proportional hazards models and their corresponding 95% Conﬁdence Intervals (95%CI). Imbalances in individual level data will be accounted for using statistical adjustment in a Mixed-Effects Cox Regression model.

Hypothesis:

This study aims to provide evidence on the effectiveness and cost-effectiveness of a individualized and protocolized nutrition intervention package for pressure injury management in home care patients. The findings could inform the development of evidence-based guidelines and recommendations for nutritional care and education in this vulnerable population, ultimately leading to improved patient outcomes and reduced healthcare costs associated with pressure injuries.

DETAILED DESCRIPTION:
Intervention:

* Individualized nutritional intervention
* receive an educational pamphlet on nutritional and wound care for patient/family based on the "The European Pressure Ulcer Advisory Panel, the National Pressure Injury Advisory Panel, and the Pan Pacific Pressure Injury Alliance Prevention and Treatment of Pressure Ulcers/Injuries: 2019 Clinical Practice Guideline", with an in-depth explanation by trained nursing staff and research dietitian.
* reinforcement of nutritional education (adequate calories/ protein/fluid intake, and compliance to consumption of supplements) by nurses on visits without dietitian.
* A dietetic consultation at baseline, 30 days, 60 days and 90 days of the intervention will be done by an experienced and trained dietitian on optimizing nutritional intake to meet energy/protein requirements. The dietetic consultation will be done via face-to-face home visits and/or teleconsultation (depending on patient and caregiver preference).
* additional high protein high energy (HPHE) supplementation (commercial ready-to-drink oral nutritional supplements, which are available in hospitals, pharmacies and retail outlets) prescribed for those participants who do not meet nutritional requirements (25-35kcal/kg/d and 1.2-2.0g protein/kg/d).
* a specialized nutritional supplement containing 4.5 g Arginine, 156 mg Vitamin C, 40.9 mg alpha-tocopherol equivalents (Vitamin E), 30 kcal will be administered twice a day via oral ingestion or tube feeding for 12 weeks (14 serves per week).
* adjustment of enteral feeding regimen will be made for those patients who have not seen a dietitian previously in their last hospital admission.
* Compliance to supplementation will be determined by recording the amount of leftover products by individuals / caregivers and confirmation of intake with the caregiver / family member during the dietitian or nursing visit at 30-day, 60-day and 90-day period.

Control:

* protocolized nutritional intervention
* receive an educational pamphlet on nutritional and wound care for patient/family based on the latest nursing and nutritional guidelines, with an in-depth explanation by trained nursing staff. The trained nurses will provide reinforcement of nutritional education on planned visits as per usual practice over the 90 days.
* Standard care and follow-up as per hospital care plans with dietitian/home nursing foundation calling hospital dietitian-in-charge of subject if necessary, for verbal advice as per usual practice.
* HPHE supplementation (commercial standard ready-to-drink oral nutritional supplements available in pharmacy) / dietary advice to meet nutritional requirements will be based on previous recommendations from hospital dietitian-in-charge/clinician review of subject.

Primary Outcome Measurements

1. Change in Pressure Injury Area from Baseline: Measurement of the alteration in the surface area of the identified pressure injury (PI) at time points of 30, 60, 90 days, 6 months and 1 year post-intervention.
2. Proportion of Participants with 40% or Greater Area Reduction: Calculation of the percentage of participants who exhibit a reduction in the PI area by at least 40% at the same time points.

Secondary Outcome Measurements

1. Proportion with Increased Severity in Pressure Injury Stages
2. Proportion with Complete Pressure Injury Healing
3. Proportion with Improvement in Health-Related Quality of Life (HRQOL)
4. Proportion with Nutritional Status Improvement
5. Change in HRQOL (EQ-5D-5L Utility Values and VAS)
6. Incidence of New Pressure Injury
7. Incidence of Pressure Injury Wound Infections
8. Mortality Rate
9. Unplanned Hospital Admissions and Length of Stay

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age more than or equal to 21 years, any gender).
2. Stage II, III, IV, and unstageable pressure injuries. For patients with multiple wounds, we will include all the pressure injuries (stages II and above) in the investigation.
3. Able to provide written informed consent (patient or legal guardian).
4. Be on oral and/or enteral nutritional support.

Exclusion Criteria:

1. Known palliative care individuals with a lifespan of </= 3 months,
2. Known septicaemia,
3. Poorly controlled diabetes (glycated haemoglobin level > 8.5%17),
4. Individuals on strict fluid restriction if the provision of additional oral or enteral nutrition supplements leads to excess intake, for the following conditions:

   1. Advanced renal disease not on dialysis (KDIGO [21, 22] Stage G4 with an estimared Glomerular Filtration Rate (eGFR) of 15-29 ml/min/1.73m2 and Stage G5 with an eGFR less than 15 ml/min/1.73m2
   2. Advanced decompensated alcoholic and non-alcoholic liver cirrhosis
   3. Heart failure with reduced ejection fraction requiring fluid restriction less than 800ml per day,

6. Previous (last chemotherapy or radiotherapy less than one year ago) or current neoplastic disease 7. Currently on immunosuppressive therapy, 8. Known allergy reaction to L-arginine, phenylketonuria 9. Presence of an infected wound (if it is the only pressure injury present on the participant) 10. Presence of untreated diagnosed osteomyelitis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the area of pressure injury from baseline | Baseline, 30 days, 60 days, 90 days, 6 months and 1 year
  Assessed by the change in wound area from baseline to the follow-up timepoints, measured with a 3D wound imaging device at the time of follow-up.
Percentage (%) of participants at time of follow-up with pressure injury wound area reduction of >/=40% | Baseline, 30 days, 60 days, 90 days, 6 months and 1 year
  Percentage (%) of participants at time of follow-up with wound area reduction >/= 40%, at time of follow-up versus baseline, where the number of patients with wound area reduction >/= 40% at follow-up timeframe will be determined as a percentage of total number of participants in the study group.

SECONDARY OUTCOMES:
Proportion of participants with complete wound healing of the main wound | 30 days, 60 days, 90 days, 6 months and 1 year
  Proportion of participants with complete wound healing of the main wound. Assessed by the number of participants with complete healing of a wound, determined by clinical assessment and pressure injury staging.
Proportion of participants with increased severity of pressure injury (PI stage) | 30 days, 60 days, 90 days, 6 months and 1 year
  Proportion of participants with increased severity of pressure injury (PI stage). Assessed by the number of participants with increased severity of wound at follow-up. Severity of pressure injury determined by the increase in pressure injury staging, or increase in area of wound if pressure injury staging remains the same at the follow-up time points
Proportion of participants with new wound infection | 30 days, 60 days, 90 days, 6 months and 1 year
  Proportion of participants with New wound infection. Assessed by the number of participants with a new wound infection(s) at follow-up, that is clinically diagnosed with confirmation from blood tests (e.g., C-Reactive Protein (CRP), renal and liver function tests).
Change in Health-Related Quality of Life (HRQOL) utility scores from baseline to time of follow-up. | 90 days, 6 months and 1 year
  Change in HRQOL assessed by the change in the EuroQOL 5-Dimensions 5-Levels (EQ5D-5L) utility scores at follow-up from baseline for the overall population and age categories if appropriate, where change in scores expressed as mean differences or standardised mean differences.
Change in Health-Related Quality of Life (HRQOL) Visual Analogue Scale (VAS) scores from baseline to time of follow-up. | 90 days, 6 months and 1 year
  Change in HRQOL assessed by the change in the EuroQOL 5-Dimensions 5-Levels (EQ5D-5L) Visual Analogue Scale (VAS) at follow-up from baseline for the overall population and age categories if appropriate, where change in scores expressed as mean differences or standardised mean differences.
Change in Nutritional status. | 30 days, 60 days, 90 days and 1 year
  Change in Nutritional status. Assessed using the Global Leadership Initiative on Malnutrition (GLIM) criteria, to determine the severity of malnutrition. Change in the nutritional status determined by direction of nutritional status shift from baseline to follow-up.
Change in Nutritional Intake. | 30 days and 60 days
  Change in Nutritional Intake. Assessed by the change in average of energy, protein and selected micronutrient intake derived from 3day food records.
Mortality | 30 days, 60 days, 90 days, 6 months and 1 year
  Mortality assessed by the occurrence and time-to-event of all-cause mortality during the study period.
Unplanned Hospital Admission | 30 days, 60 days, 90 days, 6 months and 1 year
  Unplanned hospital admission assessed by the occurrence and time-to-event of one or more admissions during the study period.

OTHER OUTCOMES:
Adherence to Nutrition Supplementation Intake | 30 days, 60 days and 90 days
  Adherence to nutrition supplementation assessed by the number of participants with >75% consumption of oral nutritional supplements and Arginaid, where the servings of products consumed are counted w confirmation of intake during follow-up.
Hospital Length of Stay | 1 year
  Hospital Length of Stay assessed by the number of days for each unplanned hospital admission.
Wound Depth | 30 days, 60 days, 90 days, 6 months and 1 year
  Wound Depth measured (millimeters) using sterile forceps and ruler at follow-up.
Wound Duration | 1 year
  Measured by days to complete heal for participants with complete wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Wong, MSc, Principal Investigator — SingHealth Duke NUS
Locations (1):
- Home Nursing Foundation, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz N, Posthauer ME, Cereda E, Schols JMGA, Haesler E. The Role of Nutrition for Pressure Injury Prevention and Healing: The 2019 International Clinical Practice Guideline Recommendations. Adv Skin Wound Care. 2020 Mar;33(3):123-136. doi: 10.1097/01.ASW.0000653144.90739.ad. PMID 32058438
- [Background] European Pressure Ulcer Advisory Panel, National Pressure Injury Advisory Panel, and Pan Pacific Pressure Injury Alliance, Prevention and Treatment of Pressure Ulcers/Injuries: Quick Reference Guide., E. Haesler, Editor. 2019
- [Background] Graves, N. and H. Zheng, The prevalence and incidence of chronic wounds: a literature review. Wound Practice & Research: Journal of the Australian Wound Management Association, 2014. 22(1): p. 4-12
- [Background] Goh OQ, Ganesan G, Graves N, Ng YZ, Harding K, Tan KB. Incidence of chronic wounds in Singapore, a multiethnic Asian country, between 2000 and 2017: a retrospective cohort study using a nationwide claims database. BMJ Open. 2020 Sep 25;10(9):e039411. doi: 10.1136/bmjopen-2020-039411. PMID 32978205
- [Background] Zhan C, Miller MR. Excess length of stay, charges, and mortality attributable to medical injuries during hospitalization. JAMA. 2003 Oct 8;290(14):1868-74. doi: 10.1001/jama.290.14.1868. PMID 14532315
- [Background] Lo ZJ, Lim X, Eng D, Car J, Hong Q, Yong E, Zhang L, Chandrasekar S, Tan GWL, Chan YM, Sim SC, Oei CW, Zhang X, Dharmawan A, Ng YZ, Harding K, Upton Z, Yap CW, Heng BH. Clinical and economic burden of wound care in the tropics: a 5-year institutional population health review. Int Wound J. 2020 Jun;17(3):790-803. doi: 10.1111/iwj.13333. Epub 2020 Mar 9. PMID 32149471
- [Background] Langer G, Fink A. Nutritional interventions for preventing and treating pressure ulcers. Cochrane Database Syst Rev. 2014 Jun 12;2014(6):CD003216. doi: 10.1002/14651858.CD003216.pub2. PMID 24919719
- [Background] Chaboyer W, Bucknall T, Webster J, McInnes E, Gillespie BM, Banks M, Whitty JA, Thalib L, Roberts S, Tallott M, Cullum N, Wallis M. The effect of a patient centred care bundle intervention on pressure ulcer incidence (INTACT): A cluster randomised trial. Int J Nurs Stud. 2016 Dec;64:63-71. doi: 10.1016/j.ijnurstu.2016.09.015. Epub 2016 Sep 23. PMID 27693836
- [Background] Cereda E, Klersy C, Andreola M, Pisati R, Schols JM, Caccialanza R, D'Andrea F; OligoElement Sore Trial (OEST) Study Group. Cost-effectiveness of a disease-specific oral nutritional support for pressure ulcer healing. Clin Nutr. 2017 Feb;36(1):246-252. doi: 10.1016/j.clnu.2015.11.012. Epub 2015 Dec 2. PMID 26703983
- [Background] Cereda E, Klersy C, Serioli M, Crespi A, D'Andrea F; OligoElement Sore Trial Study Group. A nutritional formula enriched with arginine, zinc, and antioxidants for the healing of pressure ulcers: a randomized trial. Ann Intern Med. 2015 Feb 3;162(3):167-74. doi: 10.7326/M14-0696. PMID 25643304
- [Background] Wong A, Chew A, Wang CM, Ong L, Zhang SH, Young S. The use of a specialised amino acid mixture for pressure ulcers: a placebo-controlled trial. J Wound Care. 2014 May;23(5):259-60, 262-4, 266-9. doi: 10.12968/jowc.2014.23.5.259. PMID 24810310
- [Background] Wong A, Goh G, Banks MD, Bauer JD. Economic Evaluation of Nutrition Support in the Prevention and Treatment of Pressure Ulcers in Acute and Chronic Care Settings: A Systematic Review. JPEN J Parenter Enteral Nutr. 2019 Mar;43(3):376-400. doi: 10.1002/jpen.1431. Epub 2018 Sep 12. PMID 30207386
- [Background] Husereau D, Drummond M, Augustovski F, de Bekker-Grob E, Briggs AH, Carswell C, Caulley L, Chaiyakunapruk N, Greenberg D, Loder E, Mauskopf J, Mullins CD, Petrou S, Pwu RF, Staniszewska S; CHEERS 2022 ISPOR Good Research Practices Task Force. Consolidated Health Economic Evaluation Reporting Standards 2022 (CHEERS 2022) Statement: Updated Reporting Guidance for Health Economic Evaluations. Value Health. 2022 Jan;25(1):3-9. doi: 10.1016/j.jval.2021.11.1351. PMID 35031096
- [Background] Sanders GD, Neumann PJ, Basu A, Brock DW, Feeny D, Krahn M, Kuntz KM, Meltzer DO, Owens DK, Prosser LA, Salomon JA, Sculpher MJ, Trikalinos TA, Russell LB, Siegel JE, Ganiats TG. Recommendations for Conduct, Methodological Practices, and Reporting of Cost-effectiveness Analyses: Second Panel on Cost-Effectiveness in Health and Medicine. JAMA. 2016 Sep 13;316(10):1093-103. doi: 10.1001/jama.2016.12195. PMID 27623463